CLINICAL TRIAL: NCT06965946
Title: Effectiveness of Combining Intermittent Hypoxia-Hyperoxia and Conventional Physical Therapy for Patients With Knee Osteoarthritis: A Randomized Controlled Trial
Brief Title: Intermittent Hypoxia-Hyperoxia Combined With Physical Therapy for Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Collaborators: Rehman Medical Institute - RMI (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMU/DIR/CTU/2025/002
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Osteo Arthritis Knee
Keywords: Knee Osteoarthritis; Intermittent Hypoxia; Hypoxic-Hyperoxic Therapy; Rehabilitation; Functional Mobility
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: This is a two-arm parallel-group randomized controlled trial. Participants will be randomly assigned to either the experimental group receiving intermittent hypoxia-hyperoxia therapy along with conventional physical therapy or to the control group receiving conventional physical therapy with normoxic air. Both groups will receive 12 treatment sessions over four weeks.
Who Masked: Participant, Outcomes Assessor
Masking Description: This study is double blind. Both participants and outcome assessors are blinded to group allocation. Randomization is conducted via OpenEpi, and intervention/control sessions are administered with controlled oxygen levels, but the appearance and procedures are standardized to maintain blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Hypoxia-Hyperoxia + Conventional Therapy (Experimental): Participants in this group will receive Intermittent Hypoxia-Hyperoxia Therapy (IHHT) administered using a hypoxia generator. Each session will include 4 cycles of 5 minutes of hypoxia (13-15% O₂) followed by 2 minutes of hyperoxia (40% O₂). This therapy will be provided before each conventional physical therapy session. A total of 12 sessions (3 per week for 4 weeks) will be administered. Conventional therapy will follow the current best practices used by physical therapists in tertiary care hospitals in Peshawar.
  Interventions: Procedure: Intermittent Hypoxia-Hyperoxia Therapy (IHHT); Procedure: Conventional Physical Therapy
- Conventional Therapy with Normoxic Air (Active Comparator): Participants in this group will receive only conventional physical therapy along with normoxic air (19.8% O₂) exposure using the same device setup to maintain blinding. They will receive 4 sessions of normoxia (5 minutes) followed by 2 minutes of normoxia as a placebo for IHHT. This will also be done prior to each of the 12 physical therapy sessions (3 per week for 4 weeks).
  Interventions: Procedure: Conventional Physical Therapy; Procedure: Normoxic Air Placebo

INTERVENTIONS:
Procedure: Intermittent Hypoxia-Hyperoxia Therapy (IHHT) — Participants receive 4 cycles per session of 5 minutes of hypoxia (13-15% O₂) followed by 2 minutes of hyperoxia (40% O₂) using a hypoxia generator (Olive OLV 10H). Sessions are delivered before each conventional physical therapy session, 3 times per week for 4 weeks (total 12 sessions). Participants are monitored for heart rate, blood pressure, and oxygen saturation throughout the intervention.
  Other Names: Olive OLV 10H Hypoxia Generator
  Arms: Intermittent Hypoxia-Hyperoxia + Conventional Therapy
Procedure: Conventional Physical Therapy — Participants receive individualized conventional physical therapy for knee osteoarthritis based on current clinical practices in tertiary hospitals of Peshawar. Therapy is delivered 3 times per week for 4 weeks (total 12 sessions) and includes strength training, mobility exercises, and patient education.
Procedure: Normoxic Air Placebo — Participants in the control group inhale normoxic air (19.8% O₂) using the same Olive OLV 10H hypoxia generator to maintain blinding. Each session consists of 4 cycles of 5 minutes of normoxia followed by 2 minutes of normoxia, simulating the timing of hypoxia-hyperoxia therapy. Sessions are administered prior to conventional physical therapy, 3 times per week for 4 weeks (total 12 sessions). Patients are monitored for vital signs throughout.
  Arms: Conventional Therapy with Normoxic Air

SUMMARY:
This randomized controlled trial aims to evaluate the effectiveness of combining intermittent hypoxia-hyperoxia therapy (IHHT) with conventional physical therapy in improving pain, function, gait, balance, and general health among patients with knee osteoarthritis. The study will be conducted at the Physical Therapy Department of Rehman Medical Institute, Peshawar, Pakistan, over a period of one year.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a prevalent chronic condition that leads to joint pain, stiffness, and impaired mobility, particularly among middle-aged and elderly populations. In Pakistan, knee OA is common and significantly impacts quality of life. Existing treatments are largely symptomatic and often insufficient, especially in resource-constrained settings.

Intermittent hypoxia-hyperoxia training (IHHT), involving alternating periods of low (13-15%) and high (40%) oxygen concentrations, has shown promise in improving physical and psychological outcomes in musculoskeletal disorders. However, evidence regarding its efficacy in knee OA is scarce, especially in low- and middle-income countries.

This trial seeks to explore whether the combination of IHHT and conventional physical therapy leads to superior improvements in clinical outcomes compared to conventional therapy alone. Participants will undergo 12 treatment sessions over 4 weeks. The primary outcome measures include pain (NPRS), function (KOOS), balance (Timed Up and Go Test), gait (Functional Gait Assessment), and inflammatory markers (CRP). The feasibility, safety, and effectiveness of this novel intervention will also be evaluated.

The study design includes assessor and participant blinding and uses rigorous methods including pre- and post-intervention assessments and statistical analysis with SPSS. Findings from this study may inform future guidelines for non-pharmacological, low-cost interventions for knee OA rehabilitation in similar contexts.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 45 and above.
* Participants (both male and female) with knee pain for 3 months or more with any three of the following six items: age of 50 years or more, crepitations, enlarged bone, no palpable warmth, morning stiffness for less than 30 minutes, and bony tenderness.
* Patients who can walk and have a minimum score of 4 on the Numeric Pain Rating Scale.
* Participants who have intact cognition with a score of 24 and above on Mini Mini- Mental State examination.
* Participants able to walk independently for at least 45 meters in the 6-minute walk test.
* Participants having a recent X-ray (done within the past 3 months).

Exclusion Criteria:

* Patients with hip or knee arthroplasty.
* Participants with above or below knee surgery or radiating pain to the lower limb.
* Patients with history of epilepsy, pregnancy
* Diagnosed neurological condition that affects lower-limb strength or walk (e.g., stroke/ basal ganglia dysfunction/ trauma)
* Patients who refused to participate in the study or to be randomly allocated.
* Patients receiving steroids or any medicine other than that prescribed by the screening orthopaedic surgeon.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Pain Reduction | Baseline and 4 weeks (12 sessions of therapy)
  Measured on the Numeric Pain Rating Scale (NPRS), which has levels ranging from 0 to 10 in severity. 0 indicates no pain, and 10 indicates severe pain. The scale is divided into 3 categories. 1-3 indicates mild pain, 4-6 indicates moderate pain, and 7-10 indicates severe pain.
Functional Status - KOOS Activities of Daily Living Subscale | Baseline and 4 weeks
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) will be used to assess pain, recreation and quality of life, symptoms and stiffness, ADL and functional sports. The scores of each category will be calculated and converted to percentages (100%). 0-39% will indicate severe condition, 40- 59% will indicate moderate condition, 60-79% will indicate mild condition, and 80-100% will indicate no dysfunction.
Inflammatory Marker - C-Reactive Protein (CRP) | Baseline and 4 weeks
  Change in serum CRP levels measured through a blood sample as a biomarker of osteoarthritis-related inflammation. CRP levels will be taken on a continuous scale.
Balance - Timed Up and Go Test (TUG) | Baseline and 4 weeks
  Time taken (in seconds) to rise from a chair, walk 3 meters, turn, walk back, and sit down using a stop watch. A time of < or equal to 10 seconds will be considered normal, 11-20 seconds indicates good mobility with functional indipendence. > or equal to 20 seconds indicates that person needs assistance outside, 30 seconds or more indicates that person is prone to fall. MCID for time up and Go test is 2.1 seconds.

SECONDARY OUTCOMES:
Gait Performance - Functional Gait Assessment (FGA) Score | Baseline and 4 weeks
  Evaluation of gait performance and stability using the FGA scale. Normal (score of 3) performances will be walking a distance of 6 meters in less than 5.5 seconds with no assistive device and no evidence of imbalance, a normal gait pattern, and not deviating more than 6 inches out of 12 12-inch walkway width. Mild impairment (score of 2) will be recorded when a person walks 6 meters with the use of an assistive device at a slower speed and mild gait deviation (15.24-25.4 cm) outside 12 12-inch walkway. Participants will be scored 1, moderate impairment, if they walk with a slower speed, abnormal gait pattern, evidence of imbalance, deviates 10-15 inches outside 12 12-inch walkway width. Participants will be said to have severe impairment, score of 0, if they can not walk 6 meters (20 feet) without assistance, severe gait deviations or imbalance, deviates greater than 15 inches outside 12 12-inch walkway width or will not attempt the task.
Functional mobility - 6-Minute Walk Test (6MWT) | Baseline and 4 weeks
  Distance (in meters) covered during a 6-minute walk test to assess aerobic capacity and endurance. Normal score ranges from 400-700 meters. The participants will be asked to walk for 6 minutes, and the distance covered will be noted. The MCID for the 6-minute walk test is 45 meters.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Rida Shabbir, PhD, Principal Investigator — Institute of Physical Medicine and Rehabilitation, Khyber Medical University Peshawar; Dr Haider Darain, PhD, Principal Investigator — Institute of Physical Medicine and Rehabilitation, Khyber Medical University Peshawar; Dr Aatik Arsh, PhD, Principal Investigator — Institute of Physical Medicine and Rehabilitation, Khyber Medical University Peshawar
Locations (1):
- Rehman Medical Institute, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results reported in this trial will be made available to researchers upon reasonable request. This includes outcome measures such as pain scores, gait and balance assessments, CRP levels, and KOOS subscale results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be made available beginning 6 months after publication of the trial results and will remain available for 5 years.
Access Criteria: Requests must be submitted to the principal investigator and will be reviewed by the institutional research committee. Access will be granted for scientifically sound proposals that align with the scope of the original study. A data use agreement will be required.

REFERENCES:
- [Background] Mohd Yunus MH, Lee Y, Nordin A, Chua KH, Bt Hj Idrus R. Remodeling Osteoarthritic Articular Cartilage under Hypoxic Conditions. Int J Mol Sci. 2022 May 11;23(10):5356. doi: 10.3390/ijms23105356. PMID 35628163
- [Background] Cui A, Li H, Wang D, Zhong J, Chen Y, Lu H. Global, regional prevalence, incidence and risk factors of knee osteoarthritis in population-based studies. EClinicalMedicine. 2020 Nov 26;29-30:100587. doi: 10.1016/j.eclinm.2020.100587. eCollection 2020 Dec. PMID 34505846
- [Background] Katz JN, Arant KR, Loeser RF. Diagnosis and Treatment of Hip and Knee Osteoarthritis: A Review. JAMA. 2021 Feb 9;325(6):568-578. doi: 10.1001/jama.2020.22171. PMID 33560326
- [Background] Rahimi F, Sadeghisani M, Karimzadeh A. Efficacy of transcranial direct current stimulation in patients with knee osteoarthritis: A systematic review. Neurophysiol Clin. 2023 Dec;53(6):102918. doi: 10.1016/j.neucli.2023.102918. Epub 2023 Nov 8. PMID 37944293
- [Background] Benderdour M, Martel-Pelletier J, Pelletier JP, Kapoor M, Zunzunegui MV, Fahmi H. Cellular Aging, Senescence and Autophagy Processes in Osteoarthritis. Curr Aging Sci. 2015;8(2):147-57. doi: 10.2174/1874609808666150727111530. PMID 26212056
- [Background] Chang WJ, Bennell KL, Hodges PW, Hinman RS, Young CL, Buscemi V, Liston MB, Schabrun SM. Addition of transcranial direct current stimulation to quadriceps strengthening exercise in knee osteoarthritis: A pilot randomised controlled trial. PLoS One. 2017 Jun 30;12(6):e0180328. doi: 10.1371/journal.pone.0180328. eCollection 2017. PMID 28665989
- [Background] Azizi S, Rezasoltani Z, Najafi S, Mohebi B, Tabatabaee SM, Dadarkhah A. Transcranial direct current stimulation for knee osteoarthritis: a single-blind randomized sham-controlled trial. Neurophysiol Clin. 2021 Aug;51(4):329-338. doi: 10.1016/j.neucli.2020.12.002. Epub 2020 Dec 13. PMID 33323306